CLINICAL TRIAL: NCT02503202
Title: A Phase III, Randomized, Placebo-Controlled, Clinical Trial to Study the Safety and Immunogenicity of Three Consistency Lots and a High Dose Lot of rVSV-ZEBOV-GP (V920 Ebola Vaccine) in Healthy Adults
Brief Title: Evaluation of the Safety and Immunogenicity of Three Consistency Lots and a High-Dose Lot of rVSV-ZEBOV-GP (V920 Ebola Vaccine) in Healthy Adults (V920-012)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V920-012; 2015-001658-14 (EudraCT Number); V920-012 (Other: Merck Protocol Number)
Record Dates: First submitted 2015-07-17; First posted 2015-07-20 (Estimated); Results first posted 2018-10-12 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Prevention of Ebola Infection

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- V920 Consistency Lot A (Experimental): Participants received a 1.0 mL intramuscular injection of V920 on Day 1
  Interventions: Biological: V920 Consistency Lot A
- V920 Consistency Lot B (Experimental): Participants received a 1.0 mL intramuscular injection of V920 on Day 1
  Interventions: Biological: V920 Consistency Lot B
- V920 Consistency Lot C (Experimental): Participants received a 1.0 mL intramuscular injection of V920 on Day 1
  Interventions: Biological: V920 Consistency Lot C
- V920 High-dose Lot (Experimental): Participants received a 1.0 mL intramuscular injection of V920 on Day 1
  Interventions: Biological: V920 High-dose Lot
- Placebo to V920 (Placebo Comparator): Participants received a 1.0 mL intramuscular injection of placebo on Day 1
  Interventions: Biological: Placebo to V920

INTERVENTIONS:
Biological: V920 Consistency Lot A — V920 (rVSV-ZEBOV-GP) Ebola Zaire vaccine consistency Lot A, live, attenuated, sterile solution for intramuscular injection
  Arms: V920 Consistency Lot A
Biological: V920 Consistency Lot B — V920 (rVSV-ZEBOV-GP) Ebola Zaire vaccine consistency Lot B, live, attenuated, sterile solution for intramuscular injection
  Arms: V920 Consistency Lot B
Biological: V920 Consistency Lot C — V920 (rVSV-ZEBOV-GP) Ebola Zaire vaccine consistency Lot C, live, attenuated, sterile solution for intramuscular injection
  Arms: V920 Consistency Lot C
Biological: V920 High-dose Lot — V920 (rVSV-ZEBOV-GP) Ebola Zaire vaccine high-dose lot, live, attenuated, sterile solution for intramuscular injection
  Arms: V920 High-dose Lot
Biological: Placebo to V920 — Sodium chloride 0.9%, sterile solution for intramuscular injection
  Arms: Placebo to V920

SUMMARY:
The study evaluated the safety and immunogenicity of 3 consistency lots and a high-dose lot of rVSV-ZEBOV-GP (V920 Ebola Vaccine) in healthy adults. The primary purpose of this study was to demonstrate consistency in the immune responses of participants receiving 3 separate lots of V920 through 28 days postvaccination. In addition to the 3 lot groups, a high-dose group and a placebo group were studied. A subset of participants representative of all treatment groups continued through 24 months postvaccination in the extension study for the evaluation of long-term safety. The primary hypothesis states that the geometric mean titer of anti-Zaire ebolavirus envelope (ZEBOV) glycoprotein antibody at 28 days postvaccination is equivalent across the three consistency lots.

ELIGIBILITY:
Inclusion Criteria:

* Not of reproductive potential, or of reproductive potential and agrees to avoid becoming pregnant or impregnating a partner for 2 months following study vaccination.

Exclusion Criteria:

* Is currently participating in or has participated in an interventional clinical trial with an investigational compound or device within 90 days of participation in this trial.
* Has previously been randomized in another clinical trial and received V920 or any other Ebola vaccine.
* Has been exposed to Ebola virus at any time prior to study entry.
* Is pregnant or breastfeeding or plans to conceive within 2 months following study vaccination.
* Has direct household exposure to a pregnant or lactating woman at the time of participation in this trial.
* Has had a fever (≥100.5ºF/38.0ºC) within 48 hours prior to study entry.
* Has received systemic corticosteroids (equivalent of ≥2 mg/kg total daily dose of prednisone or ≥20 mg/day for persons weighing >10 kg) for ≥14 consecutive days and has not completed treatment at least 30 days prior to study entry.
* Has received systemic corticosteroids exceeding physiologic replacement doses (~5 mg/day prednisone equivalent) within 14 days prior to study entry.
* Has received any live virus vaccine within 30 days prior to study entry or any other (nonlive virus) vaccine within 14 days prior to study entry.
* Has known or suspected impairment of immunological function (e.g., HIV positive).
* Has direct household exposure to a person with known or suspected impairment of immunological function (e.g., HIV positive).
* Has a clinically significant history of intravenous (IV) drug abuse within 12 months prior to study entry.
* Has a known allergy/sensitivity or contraindication to investigational product(s) or its/their excipients (e.g., albumin).
* Has a history of malignancy <=5 years prior to study entry except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
* Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling or child) who is investigational site or sponsor staff directly involved with this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1197 (Actual)
Dates: Start 2015-08-17 (Actual); Primary Completion 2016-05-02 (Actual); Study Completion 2017-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Halperin SA, Arribas JR, Rupp R, Andrews CP, Chu L, Das R, Simon JK, Onorato MT, Liu K, Martin J, Helmond FA; V920-012 Study Team. Six-Month Safety Data of Recombinant Vesicular Stomatitis Virus-Zaire Ebola Virus Envelope Glycoprotein Vaccine in a Phase 3 Double-Blind, Placebo-Controlled Randomized Study in Healthy Adults. J Infect Dis. 2017 Jun 15;215(12):1789-1798. doi: 10.1093/infdis/jix189. PMID 28549145
- [Derived] Grant-Klein RJ, Antonello J, Nichols R, Dubey S, Simon JK. Effects of Gamma Irradiation of Human Serum Samples from rVSVDeltaG-ZEBOV-GP (V920) Ebola Virus Vaccine Recipients on Plaque-Reduction Neutralization Assays. Am J Trop Med Hyg. 2021 Mar 29;104(5):1751-1754. doi: 10.4269/ajtmh.20-1055. PMID 33782211
- [Derived] Halperin SA, Das R, Onorato MT, Liu K, Martin J, Grant-Klein RJ, Nichols R, Coller BA, Helmond FA, Simon JK; V920-012 Study Team. Immunogenicity, Lot Consistency, and Extended Safety of rVSVDeltaG-ZEBOV-GP Vaccine: A Phase 3 Randomized, Double-Blind, Placebo-Controlled Study in Healthy Adults. J Infect Dis. 2019 Aug 30;220(7):1127-1135. doi: 10.1093/infdis/jiz241. PMID 31505665
- [Derived] Coller BG, Blue J, Das R, Dubey S, Finelli L, Gupta S, Helmond F, Grant-Klein RJ, Liu K, Simon J, Troth S, VanRheenen S, Waterbury J, Wivel A, Wolf J, Heppner DG, Kemp T, Nichols R, Monath TP. Clinical development of a recombinant Ebola vaccine in the midst of an unprecedented epidemic. Vaccine. 2017 Aug 16;35(35 Pt A):4465-4469. doi: 10.1016/j.vaccine.2017.05.097. Epub 2017 Jun 21. PMID 28647166

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1261 participants were screened and 1197 were randomized.
Groups:
- V920 Consistency Lot A: Participants received a 1.0-mL intramuscular injection of V920 consistency Lot A on Day 1
- V920 Consistency Lot B: Participants received a 1.0-mL intramuscular injection of V920 consistency Lot B on Day 1
- V920 Consistency Lot C: Participants received a 1.0-mL intramuscular injection of V920 consistency Lot C on Day 1
- V920 High-dose Lot: Participants received a 1.0-mL intramuscular injection of V920 high-dose lot on Day 1
- Placebo: Participants received a 1.0-mL intramuscular injection of placebo on Day 1
Period: Base Study: Up to Month 6
Arm/Group | V920 Consistency Lot A | V920 Consistency Lot B | V920 Consistency Lot C | V920 High-dose Lot | Placebo
Started | 266 | 265 | 267 | 266 | 133
Vaccinated | 266 | 265 | 266 | 264 | 133
Completed | 248 | 253 | 252 | 255 | 130
Not Completed | 18 | 12 | 15 | 11 | 3
Not completed — Death | 1 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 11 | 8 | 10 | 5 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 6 | 3 | 4 | 4 | 1
Not completed — Randomized not vaccinated | 0 | 0 | 1 | 2 | 0
Period: Extension: Month 6 to 24
Arm/Group | V920 Consistency Lot A | V920 Consistency Lot B | V920 Consistency Lot C | V920 High-dose Lot | Placebo
Started (A subset of US participants enrolled in Extension Study) | 119 | 130 | 112 | 137 | 68
Completed | 108 | 114 | 103 | 119 | 67
Not Completed | 11 | 16 | 9 | 18 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 4 | 8 | 6 | 10 | 1
Not completed — Physician Decision | 1 | 0 | 1 | 3 | 0
Not completed — Withdrawal by Subject | 5 | 8 | 2 | 4 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | V920 Consistency Lot A | V920 Consistency Lot B | V920 Consistency Lot C | V920 High-dose Lot | Placebo | Total
Number analyzed (Participants) | 266 | 265 | 267 | 266 | 133 | 1197
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.3 (13.4) | 41.5 (12.4) | 40.9 (13.1) | 41.7 (13.4) | 41.1 (13.7) | 41.3 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 143 | 135 | 138 | 149 | 72 | 637
  Male | 123 | 130 | 129 | 117 | 61 | 560

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titer of Anti-ZEBOV Glycoprotein Antibody
Description: Serum was collected for determination of geometric mean titer (GMT) of anti-Zaire ebolavirus envelope (ZEBOV) glycoprotein antibodies using an enzyme-linked immunosorbent assay (GP-ELISA). The unit of measure is ELISA units/mL (EU/mL). The lower limit of quantification for the assay was 36.11 EU/mL.
Time Frame: Day 28 postvaccination
Population: Participants who were compliant with the protocol, received vaccination, were seronegative at Day 1, and had a serum sample collected within the acceptable day range
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | V920 Consistency Lot A | V920 Consistency Lot B | V920 Consistency Lot C | V920 High-dose Lot | Placebo
Number analyzed (Participants) | 239 | 231 | 226 | 219 | 124
EU/mL | 1183.9 [1038.7 to 1349.4] | 1266.0 [1108.2 to 1446.2] | 1346.0 [1176.6 to 1539.9] | 1291.9 [1126.9 to 1481.2] | NA [NA to NA] — Geometric Mean and CIs are <36.11 EU/mL
Statistical Analysis 1: Comparison: V920 Consistency Lot A vs V920 Consistency Lot B; Test type: Equivalence — Lot consistency requires the 95% confidence interval of the GMT ratio of >0.5 and ≤2.0 for the primary analysis and >0.67 and ≤1.5 for the secondary analysis; p < 0.001, ANOVA — Primary analysis: a p-value <0.025 supported the conclusion of equivalence. If equivalence was established for the 3 pairwise comparisons, the lots would be considered to be consistent; GMT ratio (Lot A / Lot B) = 0.94, 95% CI 2-sided [0.77 to 1.14]
Statistical Analysis 2: Comparison: V920 Consistency Lot A vs V920 Consistency Lot C; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]; GMT ratio (Lot A / Lot C) = 0.88, 95% CI 2-sided [0.71 to 1.09]
Statistical Analysis 3: Comparison: V920 Consistency Lot B vs V920 Consistency Lot C; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]; GMT ratio (Lot B / Lot C) = 0.94, 95% CI 2-sided [0.77 to 1.15]

2. Primary Outcome: Percentage of Participants Reporting Serious Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study vaccine or protocol-specified procedure, whether or not considered related to the study vaccine or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the study vaccine or protocol-specified procedure is also an adverse event. A serious AE (SAE) is an AE that results in death, is life threatening, results in persistent or significant disability or incapacity, results in or prolongs a hospitalization, is a congenital anomaly or birth defect, is any other important medical event, is a cancer, or is associated with an overdose.
Time Frame: Up to Month 6 postvaccination
Population: Randomized participants who received vaccination and had follow-up data for the outcome measure
Measure: Number; unit: Percentage of participants
Arm/Group | V920 Consistency Lot A | V920 Consistency Lot B | V920 Consistency Lot C | V920 High-dose Lot | Placebo
Number analyzed (Participants) | 265 | 263 | 263 | 260 | 133
Percentage of participants | 2.6 | 1.5 | 2.7 | 1.2 | 0.0
Statistical Analysis 1: Comparison: V920 Consistency Lot A vs V920 Consistency Lot B; Test type: Other; p = 0.368, Miettinen & Nurminen; Risk Difference (RD) = 1.1, 95% CI 2-sided [-1.5 to 4.0] — Risk difference is Lot A - Lot B
Statistical Analysis 2: Comparison: V920 Consistency Lot A vs V920 Consistency Lot C; Test type: Other; p = 0.989, Miettinen & Nurminen; Risk Difference (RD) = -0.0, 95% CI 2-sided [-3.1 to 3.0] — Risk difference is Lot A - Lot C
Statistical Analysis 3: Comparison: V920 Consistency Lot B vs V920 Consistency Lot C; Test type: Other; p = 0.361, Miettinen & Nurminen; Risk Difference (RD) = -1.1, 95% CI 2-sided [-4.1 to 1.5] — Risk difference is Lot B - Lot C
Statistical Analysis 4: Comparison: V920 High-dose Lot vs Placebo; Test type: Other; p = 0.214, Miettinen & Nurminen; Risk Difference (RD) = 1.2, 95% CI 2-sided [-1.7 to 3.3] — Risk difference is High-dose Lot - Placebo

3. Primary Outcome: Percentage of Participants With Injection-site Adverse Events Prompted on the Vaccination Report Card
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study vaccine or protocol-specified procedure, whether or not considered related to the study vaccine or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the study vaccine or protocol-specified procedure is also an adverse event. Injection-site AEs prompted on the Vaccination Report Card (VRC) were erythema, pain, and swelling.
Time Frame: Up to Day 5 postvaccination
Population: Randomized participants who received vaccination and had follow-up data for the outcome measure
Measure: Number; unit: Percentage of participants
Arm/Group | V920 Consistency Lot A | V920 Consistency Lot B | V920 Consistency Lot C | V920 High-dose Lot | Placebo
Number analyzed (Participants) | 265 | 263 | 263 | 260 | 133
Percentage of participants
  Injection-site erythema | 14.7 | 10.6 | 14.8 | 7.3 | 1.5
  Injection-site pain | 66.8 | 73.0 | 70.3 | 67.7 | 12.8
  Injection-site swelling | 17.7 | 13.7 | 18.3 | 16.2 | 3.0
Statistical Analysis 1: Comparison: V920 Consistency Lot A vs V920 Consistency Lot B; Injection site erythema; Test type: Other; p = 0.160, Miettinen & Nurminen; Risk Difference (RD) = 4.1, 95% CI 2-sided [-1.6 to 9.9] — Risk difference is Lot A - Lot B
Statistical Analysis 2: Comparison: V920 Consistency Lot A vs V920 Consistency Lot C; Injection site erythema; Test type: Other; p = 0.971, Miettinen & Nurminen; Risk Difference (RD) = -0.1, 95% CI 2-sided [-6.2 to 6.0] — Risk difference is Lot A - Lot C
Statistical Analysis 3: Comparison: V920 Consistency Lot B vs V920 Consistency Lot C; Injection site erythema; Test type: Other; p = 0.151, Miettinen & Nurminen; Risk Difference (RD) = -4.2, 95% CI 2-sided [-10.0 to 1.5] — Risk difference is Lot B - Lot C
Statistical Analysis 4: Comparison: V920 High-dose Lot vs Placebo; Injection site erythema; Test type: Other; p = 0.016, Miettinen & Nurminen; Risk Difference (RD) = 5.8, 95% CI 2-sided [1.4 to 9.9] — Risk difference is High-dose Lot - Placebo
Statistical Analysis 5: Comparison: V920 Consistency Lot A vs V920 Consistency Lot B; Injection site pain; Test type: Other; p = 0.120, Miettinen & Nurminen; Risk Difference (RD) = -6.2, 95% CI 2-sided [-14.0 to 1.6] — Risk difference is Lot A - Lot B
Statistical Analysis 6: Comparison: V920 Consistency Lot A vs V920 Consistency Lot C; Injection site pain; Test type: Other; p = 0.380, Miettinen & Nurminen; Risk Difference (RD) = -3.5, 94% CI 2-sided [-11.4 to 4.4] — Risk difference is Lot A - Lot C
Statistical Analysis 7: Comparison: V920 Consistency Lot B vs V920 Consistency Lot C; Injection site pain; Test type: Other; p = 0.499, Miettinen & Nurminen; Risk Difference (RD) = 2.7, 95% CI 2-sided [-5.1 to 10.4] — Risk difference is Lot B - Lot C
Statistical Analysis 8: Comparison: V920 High-dose Lot vs Placebo; Injection site pain; Test type: Other; p < 0.001, Miettinen & Nurminen; Risk Difference (RD) = 54.9, 95% CI 2-sided [46.2 to 62.3] — Risk difference is High-dose Lot - Placebo
Statistical Analysis 9: Comparison: V920 Consistency Lot A vs V920 Consistency Lot B; Injection site swelling; Test type: Other; p = 0.202, Miettinen & Nurminen; Risk Difference (RD) = 4.0, 95% CI 2-sided [-2.2 to 10.3] — Risk difference is Lot A - Lot B
Statistical Analysis 10: Comparison: V920 Consistency Lot A vs V920 Consistency Lot C; Injection site swelling; Test type: Other; p = 0.878, Miettinen & Nurminen; Risk Difference (RD) = -0.5, 95% CI 2-sided [-7.1 to 6.1] — Risk difference is Lot A - Lot C
Statistical Analysis 11: Comparison: V920 Consistency Lot B vs V920 Consistency Lot C; Injection site swelling; Test type: Other; p = 0.154, Miettinen & Nurminen; Risk Difference (RD) = -4.6, 95% CI 2-sided [-10.9 to 1.7] — Risk difference is Lot B - Lot C
Statistical Analysis 12: Comparison: V920 High-dose Lot vs Placebo; Injection site swelling; Test type: Other; p < 0.001, Miettinen & Nurminen; Risk Difference (RD) = 13.1, 95% CI 2-sided [7.4 to 18.6] — Risk difference is High-dose Lot - Placebo

4. Primary Outcome: Percentage of Participants With Elevated Maximum Temperature
Description: Participants were instructed on the VRC to take and record their oral (or oral equivalent) temperature daily from the day of vaccination through Day 42. Elevated temperature was defined as ≥38.0° C (≥100.4° F).
Time Frame: Up to Day 42 postvaccination
Population: Randomized participants who received vaccination and had follow-up data for the outcome measure
Measure: Number; unit: Percentage of participants
Arm/Group | V920 Consistency Lot A | V920 Consistency Lot B | V920 Consistency Lot C | V920 High-dose Lot | Placebo
Number analyzed (Participants) | 262 | 263 | 263 | 258 | 132
Percentage of participants | 21.4 | 16.7 | 22.4 | 32.2 | 0.8
Statistical Analysis 1: Comparison: V920 Consistency Lot A vs V920 Consistency Lot B; Test type: Other; p = 0.176, Miettinen & Nurminen; Risk Difference (RD) = 4.6, 95% CI 2-sided [-2.1 to 11.4] — Risk difference is Lot A - Lot B
Statistical Analysis 2: Comparison: V920 Consistency Lot A vs V920 Consistency Lot C; Test type: Other; p = 0.769, Miettinen & Nurminen; Risk Difference (RD) = -1.1, 95% CI 2-sided [-8.2 to 6.0] — Risk difference is Lot A - Lot C
Statistical Analysis 3: Comparison: V920 Consistency Lot B vs V920 Consistency Lot C; Test type: Other; p = 0.100, Miettinen & Nurminen; Risk Difference (RD) = -5.7, 95% CI 2-sided [-12.5 to 1.1] — Risk difference is Lot B - Lot C
Statistical Analysis 4: Comparison: V920 High-dose Lot vs Placebo; Test type: Other; p < 0.001, Miettinen & Nurminen; Risk Difference (RD) = 31.4, 95% CI 2-sided [25.6 to 37.5] — Risk difference is High-dose Lot - Placebo

5. Primary Outcome: Percentage of Participants With Arthralgia or Arthritis Adverse Events Prompted on the Vaccination Report Card
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study vaccine or protocol-specified procedure, whether or not considered related to the study vaccine or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the study vaccine or protocol-specified procedure is also an adverse event. Adverse events of arthralgia and arthritis were prompted on the VRC.
Time Frame: From Day 5 to Day 42 postvaccination
Population: Randomized participants who received vaccination and had follow-up data for the outcome measure
Measure: Number; unit: Percentage of participants
Arm/Group | V920 Consistency Lot A | V920 Consistency Lot B | V920 Consistency Lot C | V920 High-dose Lot | Placebo
Number analyzed (Participants) | 265 | 263 | 263 | 260 | 133
Percentage of participants
  Arthralgia AEs | 5.7 | 5.7 | 6.5 | 7.7 | 1.5
  Arthritis AEs | 4.5 | 3.8 | 2.7 | 3.1 | 0.0
Statistical Analysis 1: Comparison: V920 Consistency Lot A vs V920 Consistency Lot B; Arthralgia; Test type: Other; p = 0.983, Miettinen & Nurminen; Risk Difference (RD) = -0.0, 95% CI 2-sided [-4.2 to 4.1] — Risk difference is Lot A - Lot B
Statistical Analysis 2: Comparison: V920 Consistency Lot A vs V920 Consistency Lot C; Arthralgia; Test type: Other; p = 0.699, Miettinen & Nurminen; Risk Difference (RD) = -0.8, 95% CI 2-sided [-5.1 to 3.4] — Risk difference is Lot A - Lot C
Statistical Analysis 3: Comparison: V920 Consistency Lot B vs V920 Consistency Lot C; Arthralgia; Test type: Other; p = 0.716, Miettinen & Nurminen; Risk Difference (RD) = -0.8, 95% CI 2-sided [-5.1 to 3.5] — Risk difference is Lot B - Lot C
Statistical Analysis 4: Comparison: V920 High-dose Lot vs Placebo; Arthralgia; Test type: Other; p = 0.012, Miettinen & Nurminen; Risk Difference (RD) = 6.2, 95% CI 2-sided [1.8 to 10.4] — Risk difference is High-dose Lot - Placebo
Statistical Analysis 5: Comparison: V920 Consistency Lot A vs V920 Consistency Lot B; Arthritis; Test type: Other; p = 0.677, Miettinen & Nurminen; Risk Difference (RD) = 0.7, 95% CI 2-sided [-2.9 to 4.4] — Risk difference is Lot A - Lot B
Statistical Analysis 6: Comparison: V920 Consistency Lot A vs V920 Consistency Lot C; Arthritis; Test type: Other; p = 0.250, Miettinen & Nurminen; Risk Difference (RD) = 1.9, 95% CI 2-sided [-1.4 to 5.4] — Risk difference is Lot A - Lot C
Statistical Analysis 7: Comparison: V920 Consistency Lot B vs V920 Consistency Lot C; Arthritis; Test type: Other; p = 0.460, Miettinen & Nurminen; Risk Difference (RD) = 1.1, 95% CI 2-sided [-2.1 to 4.5] — Risk difference is Lot B - Lot C
Statistical Analysis 8: Comparison: V920 High-dose Lot vs Placebo; Arthritis; Test type: Other; p = 0.041, Miettinen & Nurminen; Risk Difference (RD) = 3.1, 95% CI 2-sided [0.2 to 6.0] — Risk difference is High-dose Lot - Placebo

6. Primary Outcome: Percentage of Participants With Rash Adverse Events Prompted on the Vaccination Report Card
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study vaccine or protocol-specified procedure, whether or not considered related to the study vaccine or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the study vaccine or protocol-specified procedure is also an adverse event. Rash AEs prompted on the VRC were petechial rash, purpuric rash, and vesicular-type rash.
Time Frame: Up to Day 42 postvaccination
Population: Randomized participants who received vaccination and had follow-up data for the outcome measure
Measure: Number; unit: Percentage of participants
Arm/Group | V920 Consistency Lot A | V920 Consistency Lot B | V920 Consistency Lot C | V920 High-dose Lot | Placebo
Number analyzed (Participants) | 265 | 263 | 263 | 260 | 133
Percentage of participants | 3.0 | 4.6 | 3.8 | 3.8 | 1.5
Statistical Analysis 1: Comparison: V920 Consistency Lot A vs V920 Consistency Lot B; Test type: Other; p = 0.353, Miettinen & Nurminen; Risk Difference (RD) = -1.5, 95% CI 2-sided [-5.1 to 1.9] — Risk difference is Lot A - Lot B
Statistical Analysis 2: Comparison: V920 Consistency Lot A vs V920 Consistency Lot C; Test type: Other; p = 0.620, Miettinen & Nurminen; Risk Difference (RD) = -0.8, 95% CI 2-sided [-4.2 to 2.5] — Risk difference is Lot A - Lot C
Statistical Analysis 3: Comparison: V920 Consistency Lot B vs V920 Consistency Lot C; Test type: Other; p = 0.663, Miettinen & Nurminen; Risk Difference (RD) = 0.8, 95% CI 2-sided [-2.9 to 4.5] — Risk difference is Lot B - Lot C
Statistical Analysis 4: Comparison: V920 High-dose Lot vs Placebo; Test type: Other; p = 0.202, Miettinen & Nurminen; Risk Difference (RD) = 2.3, 95% CI 2-sided [-1.8 to 5.7] — Risk difference is High-dose Lot - Placebo

7. Primary Outcome: Percentage of Participants With Vesicular Lesion Adverse Events Prompted on the Vaccination Report Card
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study vaccine or protocol-specified procedure, whether or not considered related to the study vaccine or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the study vaccine or protocol-specified procedure is also an adverse event. Vesicular lesion AEs prompted on the VRC included blister and rash vesicular.
Time Frame: Up to Day 42 postvaccination
Population: Randomized participants who received vaccination and had follow-up data for the outcome measure
Measure: Number; unit: Percentage of participants
Arm/Group | V920 Consistency Lot A | V920 Consistency Lot B | V920 Consistency Lot C | V920 High-dose Lot | Placebo
Number analyzed (Participants) | 265 | 263 | 263 | 260 | 133
Percentage of participants | 1.9 | 1.1 | 1.5 | 1.5 | 0.0
Statistical Analysis 1: Comparison: V920 Consistency Lot A vs V920 Consistency Lot B; Test type: Other; p = 0.483, Miettinen & Nurminen; Risk Difference (RD) = 0.7, 95% CI 2-sided [-1.6 to 3.3] — Risk difference is Lot A - Lot B
Statistical Analysis 2: Comparison: V920 Consistency Lot A vs V920 Consistency Lot C; Test type: Other; p = 0.746, Miettinen & Nurminen; Risk Difference (RD) = 0.4, 95% CI 2-sided [-2.2 to 3.0] — Risk difference is Lot A - Lot C
Statistical Analysis 3: Comparison: V920 Consistency Lot B vs V920 Consistency Lot C; Test type: Other; p = 0.704, Miettinen & Nurminen; Risk Difference (RD) = -0.4, 95% CI 2-sided [-2.8 to 2.0] — Risk difference is Lot B - Lot C
Statistical Analysis 4: Comparison: V920 High-dose Lot vs Placebo; Test type: Other; p = 0.151, Miettinen & Nurminen; Risk Difference (RD) = 1.5, 95% CI 2-sided [-1.3 to 3.9] — Risk difference is High-dose Lot - Placebo

ADVERSE EVENTS:
Time Frame: Up to Month 24
Description: The at-risk population was randomized participants who received vaccination and had follow-up safety data available.
Arm/Group | V920 Consistency Lot A | V920 Consistency Lot B | V920 Consistency Lot C | V920 High-dose Lot | Placebo
All-Cause Mortality (participants affected / at risk) | 2/265 | 1/263 | 0/263 | 0/260 | 0/133
Serious Adverse Events (participants affected / at risk) | 12/265 | 12/263 | 11/263 | 8/260 | 4/133
Other Adverse Events (participants affected / at risk) | 211/265 | 211/263 | 208/263 | 208/260 | 35/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V920 Consistency Lot A (N=265) | V920 Consistency Lot B (N=263) | V920 Consistency Lot C (N=263) | V920 High-dose Lot (N=260) | Placebo (N=133)
Conductive deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal incarcerated hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningitis aseptic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scapula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radicular pain (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Schizophrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menometrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V920 Consistency Lot A (N=265) | V920 Consistency Lot B (N=263) | V920 Consistency Lot C (N=263) | V920 High-dose Lot (N=260) | Placebo (N=133)
Nausea (Gastrointestinal disorders) | 12 (12) | 13 (13) | 15 (16) | 14 (15) | 1 (1)
Chills (General disorders) | 14 (14) | 16 (16) | 20 (20) | 27 (27) | 1 (1)
Fatigue (General disorders) | 21 (22) | 15 (15) | 9 (9) | 20 (21) | 3 (3)
Influenza like illness (General disorders) | 14 (14) | 12 (13) | 18 (19) | 9 (9) | 1 (1)
Injection site erythema (General disorders) | 39 (43) | 30 (30) | 39 (42) | 19 (23) | 2 (2)
Injection site pain (General disorders) | 179 (198) | 192 (215) | 185 (212) | 176 (192) | 18 (19)
Injection site swelling (General disorders) | 47 (51) | 36 (40) | 49 (52) | 42 (42) | 4 (4)
Pain (General disorders) | 34 (34) | 23 (23) | 29 (30) | 32 (33) | 2 (2)
Pyrexia (General disorders) | 58 (66) | 47 (47) | 63 (70) | 76 (83) | 1 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 47 (72) | 41 (74) | 50 (75) | 53 (79) | 4 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 17 (19) | 11 (13) | 12 (12) | 23 (23) | 1 (1)
Headache (Nervous system disorders) | 61 (72) | 51 (56) | 55 (68) | 67 (83) | 15 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.